CLINICAL TRIAL: NCT01567059
Title: A Phase II Study of Tosedostat in Combination With Either Cytarabine or Decitabine in Newly Diagnosed AML or High-Risk MDS
Brief Title: Tosedostat in Combination With Cytarabine or Decitabine in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2566.00; NCI-2012-00274 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities | interventions — tosedostat; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (tosedostat and cytarabine) (Experimental): Patients receive tosedostat PO QD on days 1-35 and cytarabine IV on days 1-5.
  Interventions: Drug: tosedostat; Drug: cytarabine
- Arm II (tosedostat and decitabine) (Experimental): Patients receive tosedostat PO QD on days 1-35 and decitabine IV on days 1-5.
  Interventions: Drug: tosedostat; Drug: decitabine

INTERVENTIONS:
Drug: tosedostat — Given PO
  Other Names: aminopeptidase inhibitor CHR-2797; CHR-2797
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
  Arms: Arm I (tosedostat and cytarabine)
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
  Arms: Arm II (tosedostat and decitabine)

SUMMARY:
This study examines a new oral chemotherapy drug called tosedostat, in combination with cytarabine or decitabine. Tosedostat is thought to work by decreasing the availability of amino acids (building blocks the cell needs to make proteins) in cells. It has been shown in early studies to have activity against a variety of cancers, including leukemias. Patients with acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS) with specific genetic mutations have a poorer response to chemotherapy and a higher risk of relapse after treatment. Researchers are looking to see if combinations of chemotherapy drugs may improve outcomes for patients that do not respond as well with the current chemotherapy regimens, without increasing the risks of treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 4 month survival and complete remission (CR) rates of tosedostat in combination with either cytarabine or decitabine in untreated acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. To assess safety and tolerability of tosedostat in combination with either cytarabine or decitabine.

II. To determine the treatment related mortality defined as death within the first 30 days of beginning treatment.

III. To estimate rates of disease-free survival (DFS) and the 1 year overall survival (OS).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive tosedostat orally (PO) once daily (QD) on days 1-35 and cytarabine intravenously (IV) on days 1-5.

ARM II: Patients receive tosedostat PO QD on days 1-35 and decitabine IV on days 1-5.

If the patient develops a significant increase in their circulating or bone marrow blast count, the subsequent cycle may be started as early as day 21 of the current cycle. In both arms, treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or partial CR (pCR) may receive 2 additional courses of treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* All adults >= 60 years of age with untreated AML or high-risk MDS (10-19% marrow blasts) including those with prior myelodysplasia (MDS)/AML, therapy-related AML, AML with trilineage dysplasia (AML-TLD), and AML with adverse cytogenetics; patients may be enrolled if they received prior treatment with hydroxyurea to control blood counts or demethylating agents specifically for the purpose of treating MDS
* Adults age 18 to 59 with untreated AML or high-risk MDS and a transplant-related mortality (TRM) score of >= 9.2; previous data suggests these people would have a 25% mortality with standard therapy, making this treatment a reasonable alternative
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2
* Serum creatinine =< 2.0 mg/dL; if serum creatinine > 2.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 50 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation
* Serum bilirubin =< 1.5 × upper limit of normal (ULN) (in the absence of Gilbert's syndrome)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 3.0 × ULN
* Alkaline phosphatase =< 2.5 × ULN
* Male subjects, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Active uncontrolled infection
* Known infection with human immunodeficiency virus (HIV)
* Medical condition, serious concurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator, could jeopardize patient safety or interfere with the objectives of the study
* Uncontrolled angina or myocardial infarction within 6 months; patients with recent myocardial infarction apparently due to medical causes unrelated to underlying cardiac abnormalities must have a cardiac consult, and be cleared to participate in the research by the cardiologist prior to initiation of treatment and may be enrolled at the discretion of the primary investigator (PI) and treating physician
* Current or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, unless a screening echocardiogram (ECHO) or multiple gate acquisition scan (MUGA) performed within 1 month prior to study screening results in a left ventricular ejection fraction (LVEF) that is >= 45% (or institutional lower limit of normal value)
* Diagnosed or treated for another malignancy within 1 year of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving CR | 4 months after beginning treatment
  Defined by Cheson et al.

CONTACTS AND LOCATIONS:
Overall Officials: John Pagel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States